CLINICAL TRIAL: NCT06129968
Title: Transforming Ovarian Cancer Diagnostic Pathways (TranSforming Ovarian caNcer diAgnosTic pAthways: A Hybrid Type 1 Effectiveness-implementation Study of a Novel Biomarker Based, Threshold Driven Pathway for Earlier Ovarian Cancer Diagnosis
Brief Title: Transforming Ovarian Cancer Diagnostic Pathways
Acronym: SONATA
Status: Recruiting | Type: Observational
Sponsor: Professor Sudha Sundar (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor-Investigator, Professor Sudha Sundar, Professor of Gynaecological Cancer, Sandwell & West Birmingham Hospitals NHS Trust
Organization: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Other Study IDs: 23/WS/0107; 23/CAG/0086 (Other: Confidential Advisory Group)
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; diagnosis; Primary care; CA125; HE4; ROMA algorithm
MeSH Terms: conditions — Ovarian Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, 41000 anticipated as some patients will have repeat tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational cohort study is to compare the diagnostic accuracy and cost effectiveness of Risk of Malignancy Algorithm (ROMA) compared with CA125 in the diagnosis of ovarian cancer in patients attending their general practitioner (GP) with symptoms that sometimes might indicate ovarian cancer. The main questions it aims to answer are: • what is the accuracy of the ROMA algorithm which uses the blood tests CA125 and Human epididymis protein 4 (HE4) compared to CA125 in diagnosing ovarian cancer, particularly early-stage ovarian cancer, in women tested for suspected ovarian cancer from primary care? • What is the cost-effectiveness of ROMA versus CA125 testing in primary care to diagnose ovarian cancer? When a participant's GP orders a CA125 blood test, the blood will also be tested for HE4 and the ROMA algorithm calculated. The diagnostic accuracy of ROMA and CA125 will be compared to see if ROMA would be a better diagnostic test for ovarian cancer when used in the primary care setting.

DETAILED DESCRIPTION:
A woman's chances of surviving 5 years after Ovarian Cancer (OC) diagnosis drops from 90% if diagnosed at Stage 1 to 15% at Stage 4. Currently, GPs use a blood test called CA125 and ultrasound scan to decide whether to refer a woman to hospital for suspected OC. CA125 misses 50% of early-stage cancers (Stage 1 and 2); both tests cause unnecessary referrals. Recently, a blood test called Human epididymis protein 4 (HE4) in combination with CA125 in a formula called ROMA (Risk of Malignancy Algorithm) has been developed. ROMA is used by doctors in the US and Europe to guide referrals and recommended by the American College of Obstetrics and Gynaecology. A large Cochrane systematic review of 30,000+ patients across 50 papers shows ROMA detects more cancers at earlier stage than a combination of CA125 and ultrasound. All included studies were conducted in hospital where OC rates are high, however a model at 3% OC rate shows that ROMA is superior. Before the test can be introduced in NHS, it is necessary to confirm this evidence in a large primary care study and establish cost effectiveness. The wider NHS cancer programme funded SONATA project evaluates an integrated pathway from community to cancer specialists using ROMA. It includes National Health Service (NHS) pilots in primary and secondary care to establish how practice can be supported to change, evaluates facilitators and barriers to change as well as a community campaign to promote OC awareness. This study is one component of the SONATA project. In it, two large NHS labs will additionally test 41,000 blood samples from women whose GPs requested CA125 testing for suspected OC with ROMA to accurately identify the number of patients who can be detected earlier. This will enable the investigators to establish cost effectiveness of ROMA and definitive data on accuracy in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting to primary care with suspected ovarian cancer who are tested for the biomarker CA125 according to current standards of care for investigation of CA125 in the primary care setting.

Exclusion Criteria:

* Patients presenting to primary care who do not have potential symptoms of ovarian cancer.
* Women with symptoms sometimes associated with ovarian cancer not tested for ovarian cancer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Women presenting to primary care with suspected ovarian cancer who are tested for the biomarker CA125 according to current standards of care for investigation of CA125 in the primary care setting.
  * All samples requested by GPs for testing with CA125 in women in two large labs, Black Country Pathology Wervices and South Tyne and Wear labs, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 34000 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ROMA versus CA125 in early stage ovarian cancer | 12 months
  Cancer diagnoses will be identified from hospital gynaecological oncology centre multidisciplinary team databases.
Specificity of ROMA versus CA125 in early stage ovarian cancer | 12 months
  Cancer diagnoses will be identified from hospital gynaecological oncology centre multidisciplinary team databases.

SECONDARY OUTCOMES:
Sensitivity of ROMA versus CA125 in all stages of ovarian cancer | 12 months
  Cancer diagnoses will be identified from hospital gynaecological oncology centre multidisciplinary team databases.
Specificity of ROMA versus CA125 in all stages of ovarian cancer | 12 months
  Cancer diagnoses will be identified from hospital gynaecological oncology centre multidisciplinary team databases.
Incremental Cost Effectiveness Ratio (ICER) of ROMA versus CA125 | 12 months
  Derived from a model-based cost consequence analysis from an NHS and Personal Social Services perspective comparing the new primary care diagnostic pathway using ROMA to the standard primary care pathway of CA125 followed by ultrasound.

OTHER OUTCOMES:
Number of health care visits | 12 months
  As identified from hospital gynaecological oncology centre multidisciplinary team databases.
Rate of Emergency Hospital admissions | 12 months
  As identified from hospital gynaecological oncology centre multidisciplinary team databases.
Cancer stage | 12 months
  FIGO stage identified from hospital gynaecological oncology centre multidisciplinary team databases.
% of each treatment modality (surgical resection and chemotherapy, chemotherapy alone, surgical resection alone, or other) | 12 months
  As identified from hospital gynaecological oncology centre multidisciplinary team databases.
Survival | 12 months
  Calculated from date of death or of last point of contact and from diagnosis date recorded in hospital gynaecological oncology centre multidisciplinary team databases.

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Sundar, Principal Investigator — University of Birmingham/Sandwell and West Birmingham NHS Trust
Locations (3):
- United Kingdom (3):
  - Sandwell and West Birmingham NHS TRUST, Birmingham
  - Gateshead Health NHS Foundation Trust, Gateshead
  - The Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No